CLINICAL TRIAL: NCT05160818
Title: Hypofractionated Stereotactic Radiotherapy Versus Single Fraction Stereotactic Radiosurgery to the Resection Cavity of Brain Metastases After Surgical Resection - A Prospective, Randomized, Controlled, Monocentric Phase III Trial
Brief Title: Hypofractionated Versus Single Fraction Stereotactic Adjuvant Radiotherapy to the Resection Cavity of Brain Metastases
Acronym: SATURNUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Stephanie Combs, Univ.-Prof. Dr. med. Stephanie E. Combs, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RadOnc MRI TUM - 2
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Brain Metastases; Resection Cavity
Keywords: Brain Metastases; Resection Cavity; Radiotherapy; Stereotactic Irradiation; Gamma Knife
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: 1:1 Parallel Assignment
Masking Description: The affiliation to the treatment arm will not be blinded to anyone except the study neuroradiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: HSFRT (Active Comparator): Hypofractionated stereotactic radiotherapy to the resection cavity, dose prescription: 6-7 x 5 Gy
  Interventions: Radiation: Hypofractionated stereotactic radiotherapy (HFSRT) versus single fraction stereotactic radiotherapy radiosurgery (SRS)
- Arm B: SRS (Active Comparator): Single fraction stereotactic radiotherapy to the resection cavity, dose prescription: 1 x 12-20 Gy
  Interventions: Radiation: Hypofractionated stereotactic radiotherapy (HFSRT) versus single fraction stereotactic radiotherapy radiosurgery (SRS)

INTERVENTIONS:
Radiation: Hypofractionated stereotactic radiotherapy (HFSRT) versus single fraction stereotactic radiotherapy radiosurgery (SRS) — intervention description see above

SUMMARY:
This prospective, randomized, controlled, monocentric clinical phase III study focuses on stereotactic irradiation of resection cavities of brain metastases after surgical resection and seeks to demonstrate the superiority of fractionated irradiation schemes in terms of local control.

DETAILED DESCRIPTION:
There is a growing scientific focus on single fraction stereotactic (SRS) and hypofractionated stereotactic irradiation (HFSRT) after surgical resection of brain metastasis and its use is more frequently recommended in international guidelines. Despite intensive research, the optimal fractionation scheme and dose prescription for adjuvant irradiation of the resection cavity remains unclear.

Based on our own institutional data [Cit.1] and a recently published metaanalysis [Cit.2], we hypothesize that local control (LC) after HFSRT is superior compared to SRS in terms of LC. To evaluate the hypothesis in a prospective, randomized, controlled setting we designed the SATURNUS study.

A total of 126 patients will be randomized 1:1 to either HFSRT (dose 6-7 x 5 Gy) or SRS (dose 1 x 12-20 Gy). If further unresected brain metastases are present, they will be treated with SRS (1 x 14 - 22 Gy). Irradiation is carried out with a Gamma Knife or a Linear Accelerator. In line with current clinical practice, the choice of positioning method for SRS with the Gamma Knife (mask or stereotactic frame) is left to the patient. In the case of SRS with the Linear Accelerator or HFSRT, fixation is done with a mask as technically not otherwise feasible. Follow-up-MRI will be at least carried out 6 weeks and 3, 6, 9 and 12 months after treatment. Primary endpoint of the study is local control (LC) at the irradiated resection cavity after 12 months. Locoregional control (LRC) and overall survival (OS) as well as salvage-treatments, irradiation-associated toxicities (especially rate of radionecrosis) and quality-of-life parameters are investigated as secondary endpoints.

To the best of our knowledge, the SATURNUS study is the only randomized phase III study comparing different techniques of postoperative stereotactic radiotherapy after resection of brain metastases adequately powered to detect a superiority of HSFRT regarding LC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor disease
* One to three resected brain metastases
* Consent to perform adjuvant irradiation by an interdisciplinary tumor board
* Completed wound healing
* Resection within the last six weeks at the time of study inclusion
* Diameter of the resection cavity ≤ 4 cm (on Planning MRI)
* Age > 18 years
* KPS > 60%
* Adequate contraceptive measures for fertile women / men
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* Contraindication for repetitive contrast enhanced MRI
* Leptomeningeal disease
* Small cell histology, hematological malignancies and / or germ cell malignancies
* Previous irradiation of the brain
* Pregnant and lactating women
* Inability to understand the character and consequences of the study
* Withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Local control | 12 months after adjuvant radiotherapy
  Local control at the resected site(s)

SECONDARY OUTCOMES:
LC | 12 months after adjuvant radiotherapy
  Local control at all treated site(s)
LRC | 12 months after adjuvant radiotherapy
  Locoregional control=CNS progression free survival
OS | 12 months after adjuvant radiotherapy
  Overall survival
Salvage-free survival | 12 months after adjuvant radiotherapy
  Overall survival
Intracranial salvage therapy | 12 months after adjuvant radiotherapy
  Number and kind of intracranial salvage treatments
Pseudoprogression | up to 12 months after adjuvant radiotherapy
  Rate of pseudoprogression
Irradiation-related toxicity | up to 12 months after adjuvant radiotherapy
  according to CTCAE v4.03, especially rate of radionecrosis
QoL | up to 12 months after adjuvant radiotherapy
  Quality of life according to EORTC QLQ-C30 and EORTC QLQ-B20
Time to loss of independence | up to 12 months after adjuvant radiotherapy
  defined as decrease in Barthel index by > 20 points

CONTACTS AND LOCATIONS:
Overall Officials: Maria Waltenberger, Study Director — Technical University Munich, Germany
Locations (1):
- Dept. Radiation Oncology, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Specht HM, Kessel KA, Oechsner M, Meyer B, Zimmer C, Combs SE. HFSRT of the resection cavity in patients with brain metastases. Strahlenther Onkol. 2016 Jun;192(6):368-76. doi: 10.1007/s00066-016-0955-2. Epub 2016 Mar 10. PMID 26964777
- [Background] Akanda ZZ, Hong W, Nahavandi S, Haghighi N, Phillips C, Kok DL. Post-operative stereotactic radiosurgery following excision of brain metastases: A systematic review and meta-analysis. Radiother Oncol. 2020 Jan;142:27-35. doi: 10.1016/j.radonc.2019.08.024. Epub 2019 Sep 25. PMID 31563407
- [Derived] Waltenberger M, Bernhardt D, Diehl C, Gempt J, Meyer B, Straube C, Wiestler B, Wilkens JJ, Zimmer C, Combs SE. Hypofractionated stereotactic radiotherapy (HFSRT) versus single fraction stereotactic radiosurgery (SRS) to the resection cavity of brain metastases after surgical resection (SATURNUS): study protocol for a randomized phase III trial. BMC Cancer. 2023 Jul 29;23(1):709. doi: 10.1186/s12885-023-11202-9. PMID 37516835